CLINICAL TRIAL: NCT01594203
Title: Contribution of F18-FDG PET/CT to the Early Assessment of Pazopanib Therapy Efficacy in Advanced Soft Tissue Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0103-12-HMO
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-04

CONDITIONS: Soft Tissue Sarcoma (STS)
Keywords: Soft Tissue Sarcoma; Pazopanib; F18-FDG PET/CT
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Advanced Soft Tissue Sarcoma: patients with advanced Soft Tissue Sarcoma
  Interventions: Other: F18-FGD PET/CT

INTERVENTIONS:
Other: F18-FGD PET/CT

SUMMARY:
Soft Tissue Sarcoma (STS) is a rare tumor but can grow in different areas, for example, in 60% in limbs and about 20 % in retroperitoneum; and frequently is inoperable. Despite novel therapy in advanced cases survival is still short, approximately 12 month.

Pazopanib oral angiogenesis inhibitor was recently shown as promising drug for advanced pretreated STS.

Functional imaging especially F18-FDG PET/CT is a good modality for FDG avid tumor either for pre- / post- treatment evaluation or follow up.

Early detection of treatment response to therapy by whole body FDG PET/CT allows for change of treatment as early as possible,when the tumor is non-responsive before serious side effects appear or before depletion of body resources.

The aim of the study is to investigate the contribution of FDG PET/CT to assessment of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced Soft Tissue Sarcoma prior to pazopanib treatment

Exclusion Criteria:

* Other treatment
* FDG negative tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced Soft Tissue Sarcoma prior to pazopanib therapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-11 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Measure of extent and intensity (standardized uptake value - SUV) of disease demonstrated on PET/CT images before and after treatment. | 1 week
determination of treatment efficiency by comparison of PET data (SUV) with CT changes (cm)in 3 studies and clinical information. | 4 week

SECONDARY OUTCOMES:
prediction of treatment efficiency | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel